CLINICAL TRIAL: NCT06952062
Title: Identification and Validation of a Prediction Model for CARDIOvascular Events in Patients With Multiple COMorbidities (CARDIO-COM)
Brief Title: Identification and Validation of a Prediction Model for CARDIOvascular Events
Acronym: CARDIO-COM
Status: Active, not recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 7517
Record Dates: First submitted 2025-04-23; First posted 2025-04-30 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Cardiovascular Diseases
Keywords: Cardiovascular Diseases; Venous thromboembolism; Cancer; Bleeding; Risk Assessment Model
MeSH Terms: conditions — Cardiovascular Diseases; Venous Thromboembolism; Neoplasms; Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background: Cardiovascular risk stratification is a cornerstone of modern preventive medicine, particularly in patients with multiple comorbidities, where risk estimation is inherently complex. Existing tools such as SCORE2 and the CUORE project provide important insights into cardiovascular risk but are limited in their ability to account for the interplay of multiple coexisting conditions.

Objective: The primary aim of this prospective cohort study is to develop and validate a novel cardiovascular risk prediction model specifically tailored for patients with at least two concomitant chronic diseases. Secondary objectives include comparing the predictive performance of the new model with that of SCORE2 and the CUORE project, and quantifying the incidence of venous thromboembolism (VTE), bleeding, and overall mortality in this high-risk population.

Methods: This is a prospective, monocentric, observational cohort study with an expected duration of 144 months. Patients ≥18 years with at least two of a predefined list of chronic conditions will be recruited at the Thrombosis Unit of Fondazione Policlinico Universitario A. Gemelli IRCCS. Clinical, laboratory, and instrumental data will be collected at baseline and during annual follow-up visits, for a maximum follow-up period of 10 years. Major cardiovascular events, VTE, bleeding, and mortality will be recorded. A Fine & Gray competing risks model will be applied for risk modeling, with subsequent validation in an independent cohort. Model discrimination and calibration will be evaluated using time-dependent ROC curves and calibration plots.

Expected Outcomes: The study aims to generate a robust and clinically applicable cardiovascular risk prediction model that better reflects the complexity of patients with multimorbidity. The model is expected to improve individualized prevention strategies and optimize resource allocation in clinical practice.

Ethical Considerations: The study will be conducted in accordance with the Declaration of Helsinki and Good Clinical Practice guidelines. Informed consent will be obtained from all participants.

ELIGIBILITY:
Inclusion Criteria:

* History of at least two of the following conditions: arterial hypertension, dyslipidemia, type 2 diabetes mellitus, ischemic heart disease, heart failure with reduced or preserved ejection fraction, atrial fibrillation, cardiac valvular disease, cerebrovascular disease, obesity, chronic obstructive pulmonary disease, chronic kidney disease, neoplasia (except localized basal cell or squamous cell skin neoplasms), active or previous venous thromboembolism.
* Age greater than 18 years.
* Expression of Informed Consent.

Exclusion Criteria:

* Unable or unwilling to perform follow-up visits.
* Life expectancy < 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of patients already affected by at least two pathologies at the time of the visit, prospectively recruited at the time of the first outpatient visit at the U.O.S.D. Percorso Trombosi of the I.R.C.C.S. Fondazione Policlinico Universitario Agostino Gemelli in Rome.
Sampling Method: Non-Probability Sample
Enrollment: 2400 (Estimated)
Dates: Start 2025-04-03 (Actual); Primary Completion 2037-05-02 (Estimated); Study Completion 2037-05-02 (Estimated)

PRIMARY OUTCOMES:
Major Cardiovascular Events | 10 years
  acute coronary syndrome, coronary revascularization, stroke
Major Limbs Events | 10 years
  acute limb ischemia of the lower limbs or need for revascularization of the lower limbs
Venous Thromboembolism | 10 years
  Deep vein thrombosis of the lower limbs or Pulmonary embolism

SECONDARY OUTCOMES:
Venous thromboembolism | 10 years
  Venous thromboembolism in unusual sites (i.e., upper limb, splanchnic, cerebral, ovarian, atrial)
Bleeding | 10 years
  Major and non-major clinically relevant bleeding events
Death | 10 years
  Mortality for any cause

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Pola, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome, Italy

IPD SHARING:
Plan to Share IPD: No